CLINICAL TRIAL: NCT06656247
Title: Biobanks, Registries and National Health Records: Modelling a Networking Strategy to Foster Research and Development and to Support the Secondary Use of Data and Samples of Rare Disease Patients: Implementing Dynamic Consent for Rare Disease Patients
Brief Title: Implementing Dynamic Consent for Rare Disease Patients
Acronym: ConsDinamico
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other)
Responsible Party: Principal Investigator, Luca Sangiorgi, Director of Rare Skeletal Diseases Department, Istituto Ortopedico Rizzoli
Other Study IDs: 343/2024/Oss/IOR; PNRR-MR1-2023-12377715 (Other Grant/Funding Number: Ministero della Salute - PNRR: M6/C2_CALL2023)
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Rare Disorders
Keywords: Dynamic Consent; Rare Diseases; Digital Tool; Informed Consent; Patient Engagement
MeSH Terms: conditions — Rare Diseases; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online consenting — The design and establishment of an innovative digital tool (a software application) to implement the dynamic consent and allowing interaction among healthcare professionals and patients

SUMMARY:
The study aims to test on a cohort of rare patients a digital innovative tool to support patients/parents in the informed consent and assent process and to keep up-to-date a lawful informed and dynamic consent and to use samples and data for research purposes. This will favour their engagement in clinical studies, a step which is well known to be very demanding, particularly in the rare diseases scenario, and stimulate a bidirectional dialogue between researchers and patients/parents/legal representatives.

DETAILED DESCRIPTION:
The study is organized into three main steps. Firstly, an anonymous Consent Survey, will be prepared to collect the opinions of stakeholders engaged in the RDs on strengths and weaknesses of the process of consent and assent collection. This Survey will be conducted through SurveyMonkey or similar tools, posted on websites and social media, and made available to all stakeholders (patients, carers, healthcare professionals, patient associations). Key topics like the proper consideration of paediatric specificities due to age-dependent characteristics and patient satisfaction in terms of information received during the consent/assent process will be addressed.

The survey will comprise multiple-choice and open questions. Expectations related to the use of dynamic consent, potential disbeliefs, and tools for promoting and regulating participation into future research studies (text, video) will also be evaluated. Statistical analysis on survey results, as well as sentiment analysis, will be performed.

The second step will consist of two main activities:

A) the realization of dynamic informed consent and assent templates for the processing and management of data and samples. The templates will be drafted based on the long-standing experience of the research teams and the outcomes of the Consent Survey, along with the available literature and guidelines. They will be designed in full compliance with the GDPR as implemented by the Italian legislation. Information on patients' rights, purposes of data usage, legal basis and measures taken to implement lawfulness of data processing will be included.

B) The design and establishment of an innovative digital tool (a software application) to implement the dynamic consent and allowing interaction among healthcare professionals and patients. This tool will be designed considering multiple aspects, like Consent Survey results. Firstly, this tool will guide patients and caregivers to a rapid and easy access to their consent/assent, allowing them to have a clear picture of their consented studies and consenting preferences, to possibly modify and/or withdraw their consent. Secondly, new studies will be synthetically published on the digital tool, in order to favour the patients' engagement, with a particular attention to adolescents and young adults who are more familiar with these approaches, being digital natives. RD patients may be re-contacted to be informed about any new purposes of data and sample processing. The digital tool will allow healthcare professionals to give feedback on ongoing studies and to present results in layman's terms to patients. Finally, it will be of help in critical steps of the research process, such as re-consenting procedures for minors who reach the age of legal competency. Considering all the mentioned components, the digital tool will promote a high-level of transparency. The final positive impact expected is an improved process resulting in reduced costs for both patients and the National Health System. In fact, the integration of data from multiple sources will result in increased knowledge and dissemination of correct information directly to patients thus drastically reducing misinformation, duplicate visits, and optimizing patient enrolment.

The third step of this aim is the test and validation of the dynamic consent in a cohort of rare patients. Enrolling centers, both dealing with RD patients' consent on a daily basis, will conduct a pilot study enrolling a cohort of RD patients (min. 50 subjects) during clinical routine care. This step will comprise a satisfaction questionnaire - proposed to all participating patients and carers - with the final aim of identifying pitfalls and opportunities of this innovative consenting approach, and eventually implement the digital tool according to the collected responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by a rare disease (based on clinical or genetic findings)
* Patients with a suspect of rare disease (based on clinical or genetic findings)

Exclusion Criteria:

* All patients who do not meet the inclusion criteria will be excluded from the study

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All rare patients diagnosed or followed up at IRCCs istituto Ortopedico Rizzoli and Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Test the usability of dynamic consent in a cohort of rare patients | From platform establishment, an average of 1 year
  Collect a satisfaction questionnaire - proposed to all participating patients and carers - aiming to aim of identifying pitfalls and opportunities of this innovative consenting approach

SECONDARY OUTCOMES:
Ammeliorate the dynamic consent platform following indications received by rare patients and their carer | After completion of primary outcome, an avaerage 2 months
  The survey that will be circulated to the different stakeholders and the evaluation questionnaire that will be requested from the participants will allow us to gather opinions and feedback on what has been achieved, in order to evaluate and implement a model that corresponds to the existing panorama, and subsequently also to improve it in terms of use, in the light of the content collected.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merlec MM, Lee YK, Hong SP, In HP. A Smart Contract-Based Dynamic Consent Management System for Personal Data Usage under GDPR. Sensors (Basel). 2021 Nov 30;21(23):7994. doi: 10.3390/s21237994. PMID 34883997
- [Background] Prictor M, Lewis MA, Newson AJ, Haas M, Baba S, Kim H, Kokado M, Minari J, Molnar-Gabor F, Yamamoto B, Kaye J, Teare HJA. Dynamic Consent: An Evaluation and Reporting Framework. J Empir Res Hum Res Ethics. 2020 Jul;15(3):175-186. doi: 10.1177/1556264619887073. Epub 2019 Nov 15. PMID 31729900
- [Background] Dankar FK, Gergely M, Malin B, Badji R, Dankar SK, Shuaib K. Dynamic-informed consent: A potential solution for ethical dilemmas in population sequencing initiatives. Comput Struct Biotechnol J. 2020 Apr 2;18:913-921. doi: 10.1016/j.csbj.2020.03.027. eCollection 2020. PMID 32346464
- [Background] Grady C. Enduring and emerging challenges of informed consent. N Engl J Med. 2015 Feb 26;372(9):855-62. doi: 10.1056/NEJMra1411250. PMID 25714163
- [Background] Cocanour CS. Informed consent-It's more than a signature on a piece of paper. Am J Surg. 2017 Dec;214(6):993-997. doi: 10.1016/j.amjsurg.2017.09.015. Epub 2017 Sep 20. PMID 28974311
- See also: GDPR — https://eur-lex.europa.eu/legal-content/IT/TXT/?uri=uriserv:OJ.L_.2016.119.01.0001.01.ITA&toc=OJ:L:2016:119:TOC